CLINICAL TRIAL: NCT02196389
Title: Comparison Between 4 Different Nasal Dilators: Objective vs Subjective Parameters
Brief Title: Comparison Between 4 Different Nasal Dilators
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No contract, no costs
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S56842
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Incompetence of Nasal Valve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nozovent (Active Comparator): Nasal Dilator
  Interventions: Device: Nasal dilator Nozovent
- Nasanita (Active Comparator): Nasal Dilator
  Interventions: Device: Nasal dilator Nasanita
- Breath Right (Active Comparator): Nasal Dilator
  Interventions: Device: Nasal dilator Breath Right
- Airmax (Active Comparator): Nasal Dilator
  Interventions: Device: Nasal dilator Airmax

INTERVENTIONS:
Device: Nasal dilator Nasanita — Nasal Dilator
  Other Names: Nasanita
  Arms: Nasanita
Device: Nasal dilator Nozovent
  Arms: Nozovent
Device: Nasal dilator Breath Right
  Arms: Breath Right
Device: Nasal dilator Airmax
  Arms: Airmax

SUMMARY:
Several nasal dilators are currently commercially available, and can be applied endonasally (Airmax°, Nozovent and Nasanita°) or externally (Breath Right°). An objective comparison between these dilators has not been made so far, and would help the clinicians to advise the use of any of these dilators. From clinical experience, endonasal dilators are well supported and improve breathing better than the external dilators

DETAILED DESCRIPTION:
Several nasal dilators are currently commercially available, and can be applied endonasally (Airmax°, Nozovent and Nasanita°) or externally (Breath Right°). An objective comparison between these dilators has not been made so far,

ELIGIBILITY:
Inclusion Criteria:

Patients with nasal obstruction due to external nasal valve problems and with positive Cottle sign.

Age > 18 and < 60 years. Ability to give reliable information and written informed consent.

Exclusion Criteria:

Patients with nasal obstruction due to other endonasal anatomic deformities besides external nasal valve dysfunction.

Patients with rhinosinusitis and/or nasal polyps evaluated by nasal endoscopy. Patients with chronic lower airway disease like severe asthma, chronic obstructive pulmonary disease (COPD), bronchiectasis and/or other conditions that interfere with the generation of a reliable Peak Nasal Inspiratory Flow (PNIF) result.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

PRIMARY OUTCOMES:
Peak Nasal Inflammatory Flow | 4 weeks
  Change in Peak Nasal Inflammatory Flow between the 4 different dilators

SECONDARY OUTCOMES:
preference | 4 weeks
  Patients' preference of 2 out of 4 dilators tested at baseline for a trial period of 4 week duration.

OTHER OUTCOMES:
surgery | 4 weeks
  Patients' preference to continue to use the preferred dilator after the 4 weeks' trial period or choice to undergo surgery after one month of usage of the preferred dilator.
reasons of choice | 4 weeks
  Specific reasons for the choice of the two dilators at baseline (functional vs aesthetic) at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, Prof Dr, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium